CLINICAL TRIAL: NCT03672045
Title: Carbetocin at Elective Cesarean Deliveries: A Dose-finding Study in Women With BMI ≥ 40kg/m2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-07
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Intervention Model Description: Biased coin up-and-down design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Carbetocin 10mcg (Active Comparator): Patient is given 10 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 20mcg (Active Comparator): Patient is given 20 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 40mcg (Active Comparator): Patient is given 40 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 60mcg (Active Comparator): Patient is given 60 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 80mcg (Active Comparator): Patient is given 80 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator): Patient is given 100 mcg of carbetocin intravenously over 1 minute, immediately upon delivery of the fetal head.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — carbetocin administered IV, over 1 minute following delivery of the fetal head
  Other Names: Duratocin

SUMMARY:
Postpartum hemorrhage (PPH) due to uterine atony is a major cause of maternal morbidity and mortality. Carbetocin is a uterotonic with a superior pharmacokinetic profile to oxytocin. In a study performed at Mount Sinai Hospital, the investigators have shown that smaller doses of carbetocin (14.8 mcg) are as effective in achieving adequate uterine tone at elective cesarean section compared to the current recommended dose of 100mcg. However, this study was limited to those women with a body mass index (BMI) of <40 kg/m2. Maternal obesity has been shown to increase the risks of hemorrhage secondary to uterine atony, therefore the investigators wish to perform a dose finding study to determine the ED90 of carbetocin at caesarean section in those women with a BMI>40.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is one of the leading causes of death during childbirth and accounts for an estimated 140,000 deaths per year worldwide. The World Health Organization (WHO) recommends active management of the third stage of labor to prevent PPH, even in low risk patients. Prophylactic uterotonic drugs administered after delivery are the main element of active management of the third stage and have been demonstrated to reduce the incidence of PPH by up to 40%.

Oxytocin is the most commonly used uterotonic in North America, however it has a very short duration of action and requires a continuous infusion to achieve sustained effect, with large doses associated with adverse effects like low blood pressure, nausea, vomiting, abnormal heart rhythms and changes on ECG. Carbetocin is a synthetic oxytocin analogue. It causes uterine contraction via the same mechanism as oxytocin. Its duration of action is 4 to 7 times that of oxytocin due to an increased biological half-life in plasma and at the oxytocin receptors in the uterus. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recommended a single dose of 100 mcg of carbetocin at elective cesarean delivery to promote uterine contraction. In a study performed at Mount Sinai Hospital, the investigators have shown that smaller doses of carbetocin (14.8 mcg) are effective in achieving adequate uterine tone at elective cesarean section. However this study was limited to those women with a BMI of <40 kg/m2

The prevalence of obesity is increasing in young women and some studies have shown that obese women have higher rates of caesarean delivery compared to non-obese women. Other studies have demonstrated an increased risk of hemorrhage due to poor uterine tone in obese women. Laboratory studies show that BMI alone appears to contribute to blunted uterine muscle responses and therefore contraction responses to oxytocin in obese women. Previous dose finding studies have excluded those women with a BMI of ≥40kgm2. Therefore, the investigators wish to perform a double-blind dose finding study using the biased coin up-and-down sequential allocation technique to determine the ED90 of carbetocin at caesarean section in those women with a BMI>40.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥40kg/m2
* Elective cesarean delivery under regional anesthesia
* Gestational age ≥ 37 weeks
* No known additional risk factors for postpartum hemorrhage
* Written informed consent to participate in this study

Exclusion Criteria:

* Refusal to give written informed consent
* Allergy or hypersensitivity to carbetocin or oxytocin
* Conditions (other than high BMI) that may predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* Hepatic, renal, and vascular disease
* Use of general anesthesia prior to the administration of the study drug

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Intraoperative requirement for additional uterotonic medication | 1 hour
  A request made by the obstetrician performing the cesarean delivery for additional uterotonic medication, due to bleeding or poor uterine tone.

SECONDARY OUTCOMES:
Uterine tone 2 minutes | 2 minutes
  Uterine tone, defined as satisfactory or unsatisfactory by the obstetrician at 2 minutes after completion of the carbetocin injection.
Uterine tone 5 minutes | 5 minutes
  Uterine tone, defined as satisfactory or unsatisfactory by the obstetrician at 5 minutes after completion of the carbetocin injection.
Additional uterotonics administered | 45 minutes
  The drug, dosage and timing of any additional uterotonic medication given during surgery.
Estimated blood loss | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to surgery and 24 hours after the cesarean delivery.
Intravenous fluid administered during surgery | 2 hours
  The total volume (ml) of fluid administered from entering the operating room to skin closure.
Hypotension: systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, from drug administration until end of surgery
Tachycardia: heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, from drug administration until end of surgery
Bradycardia: heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline or a heart rate < 50bpm, from drug administration until end of surgery
Presence of ventricular tachycardia: ECG | 2 hours
  Presence of ventricular tachycardia as recorded by ECG, from drug administration until end of surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, from drug administration until end of surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, from drug administration until end of surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea and number of episodes, from drug administration until end of surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting and number of episodes, from drug administration until end of surgery
Presence of chest pain: questionnaire | 2 hours
  Any presence of chest pain, from drug administration until end of surgery, as reported by the patient
Presence of shortness of breath: questionnaire | 2 hours
  Any presence of shortness of breath, from drug administration until end of surgery, as reported by the patient
Presence of headache: questionnaire | 2 hours
  Any presence of headache, from drug administration until end of surgery, as reported by the patient
Presence of flushing: questionnaire | 2 hours
  Any presence of flushing, from drug administration until end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drew T, Balki M, Farine D, Ye XY, Downey K, Carvalho JCA. Carbetocin at elective caesarean section: a sequential allocation trial to determine the minimum effective dose in obese women. Anaesthesia. 2020 Mar;75(3):331-337. doi: 10.1111/anae.14944. Epub 2019 Dec 22. PMID 31867715